CLINICAL TRIAL: NCT05456061
Title: Effect of Aqueous-Deficient Dry Eye on Lipid Layer Thickness Measurements
Brief Title: Effect of ADDE on Tear Interferometry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Kyoung Yul Seo, Prof., Yonsei University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 4-2018-0634
Record Dates: First submitted 2022-07-03; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Tear; Dry Eye Syndromes
MeSH Terms: conditions — Lacerations; Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Participants were classified into four groups: control group (Group 1), 3% diquafosol group (Group 2), punctal plug insertion group (Group 3), and combined treatment group (Group 4).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (No Intervention): No intervention
- Group 2 (Active Comparator): 3% diquafosol eye drops 6 times / day
  Interventions: Drug: 3% diquafosol eyedrops
- Group 3 (Active Comparator): Punctal plug insertion, lower eyelid
  Interventions: Procedure: Silicone punctal plug insertion
- Group 4 (Active Comparator): 3% diquafosol eye drops 6 times / day + Punctal plug insertion, lower eyelid
  Interventions: Drug: 3% diquafosol eyedrops; Procedure: Silicone punctal plug insertion

INTERVENTIONS:
Drug: 3% diquafosol eyedrops — Diquas® (Santen, Osaka, Japan), six times per day.
  Arms: Group 2; Group 4
Procedure: Silicone punctal plug insertion — a silicone punctal occluder (Parasol® Punctal Occluder, BVI, Waltham, Massachusetts, USA), inserted into the lower eyelid
  Arms: Group 3; Group 4

SUMMARY:
Importance: Lipid layer thickness (LLT) reflects the lipid components of tear film, but is affected by the mucocutaneous components. This study investigated the therapeutic effect of the treatments for aqueous-deficient dry eye (ADDE) on LLT.

Objective: To investigate the effect of ADDE and its treatments on LLT measurements by tear interferometry.

Design, Setting, and Participants: This prospective comparative interventional study included 152 eyes from 152 patients with ADDE.

Interventions: Participants were classified into four groups: control group (Group 1), 3% diquafosol group (Group 2), punctal plug insertion group (Group 3), and combined treatment group (Group 4).

Main Outcomes and Measures: Average LLT (LLTave) was measured using a LipiView® II tear interferometer at baseline and one month after treatments.

ELIGIBILITY:
Inclusion Criteria:

1. presence of one or more subjective symptoms of DED, including eye dryness, foreign body sensation, irritation, burning, blurred vision, and pain.
2. tear meniscus height (TMH) of <200 µm for aqueous deficiency measured using Keratograph 5M® (Oculus Optikgeräte GmbH, Wetzlar, Germany).
3. evidence of corneal and/or conjunctival damage on slit-lamp biomicroscopy with fluorescein staining.

Exclusion Criteria:

1. acute and chronic ocular surface diseases that affect DED, including infection, allergy, and autoimmune disease, and that interfere with tear interferometric measurements, such as corneal opacity and pterygium, were excluded.
2. a history of the use of contact lens, known systemic diseases such as Sjögren's syndrome, Stevens-Johnson syndrome, and ocular graft-versus-host disease.
3. any medical/surgical history related to tear production and tear function except that in the study protocol were excluded.
4. Hypersecretory meibomian gland dysfunction (MGD)

   * When both eyes of a patient could be included, an eye with the lower TMH was selected.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Average LLT (LLTave) | Baseline and one month after 1 month of treatments
  LLT was measured using the LipiView® II tear interferometer (Johnson & Johnson, New Brunswick, New Jersey, USA). The tear interferometer automatically records 20-second videos reflecting the TFLL on the inferior cornea. Simultaneously, the quantified LLT is measured over time in the interferometric color unit (ICU). One ICU corresponds to approximately 1 nm of LLT. The LipiView® II interferometer provides the average, maximum, and minimum LLT values. The average LLT (LLTave) reflects the LLT value at the stable phase of the TFLL spreading or equilibrium state.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No